CLINICAL TRIAL: NCT00685074
Title: Computer-based Brief Intervention for Perinatal Drug, Alcohol, and Tobacco Abuse
Brief Title: Computer-based Brief Intervention for Perinatal Substance Abuse
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Steven J. Ondersma, Associate Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MES-III; 5R01DA021329-04 (NIH); DA021329-01
Record Dates: First submitted 2008-05-23; First posted 2008-05-28 (Estimated); Last update posted 2011-10-14 (Estimated); Status verified 2011-10

CONDITIONS: Substance Abuse
Keywords: Motivational Interview; Computer based intervention; Substance abuse; post-partum
MeSH Terms: conditions — Substance-Related Disorders | interventions — Flowering time control protein FCA, Arabidopsis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Brief computer-delivered intervention for drug use (Experimental): A single interactive computer intervention based primarily on Motivational Interviewing principles.
  Interventions: Behavioral: Computer-based Motivational Interviewing
- Time control for drug use (Placebo Comparator): An series of innocuous and therapeutically inactive computer segments.
  Interventions: Behavioral: Time control

INTERVENTIONS:
Behavioral: Computer-based Motivational Interviewing — The software includes three intervention components - pros and cons, feedback, and optional goal-setting in a fixed order.
  Other Names: Motivation Enhancement System
  Arms: Brief computer-delivered intervention for drug use
Behavioral: Time control — A series of therapeutically inactive videos and questions to (a) maintain RA blind, and (b) serve as a time control.
  Arms: Time control for drug use

SUMMARY:
The purpose of the study is to see if a brief computer program can help new mothers cut down or quit tobacco, alcohol, or drug use.

DETAILED DESCRIPTION:
The purpose of this Stage I/II intervention study (that is, Stage II for drug use and Stage I for alcohol use and smoking) is to test the efficacy of a brief, computerized motivational intervention for substance abuse among post-partum women. The study will randomly assign 350 post-partum women to either intervention or control conditions, with intervention itself taking approximately 30 minutes in the period before the participant leaves the hospital. Inclusion criteria will include post-partum status, age between 18 and 45, ability to understand spoken English, and meeting criteria for one of the three substance use groups: any illicit drug use in month prior to pregnancy, meeting T-ACE criteria for problem alcohol use, or smoking in past month. Exclusion criteria will include receipt of narcotic pain medication in the past 3 hours, no sleep since giving birth, and inability to provide informed consent (e.g., due to psychosis or other clear cognitive impairment).

Lab-based follow-up will occur at 3- and 6-months postpartum. The primary outcomes will be participant report of frequency of substance use and toxicological analyses of substance use (urinalysis and expired breath CO at 3 and 6 month follow-up, hair analysis at 6-month follow-up). Secondary outcome measures include HIV risk behaviors, receipt of treatment services, motivation to change, self-efficacy, mental health functioning, violence exposure, and consequences related to substance use.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized women in immediate post-partum period
* Self report of illicit drug use, problem alcohol use, or tobacco use in month prior to pregnancy

Exclusion Criteria:

* Frank psychosis or other cognitive impairment
* Inability to communicate in English
* No sleep since giving birth
* Recent receipt of narcotic pain medication
* Grieving over medically compromised infant

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 143 (Actual)
Dates: Start 2007-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Drug use at 3 months | 3 months
Drug use at 6 months | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Steven J. Ondersma, PhD, Principal Investigator — Wayne State University
Locations (1):
- Hutzel Women's Hospital, Detroit, Michigan, United States